CLINICAL TRIAL: NCT01244126
Title: Postoperative Analgesic and Behavioral Effects of Intranasal Fentanyl, Intravenous Morphine and Intramuscular Morphine in Pediatric Patients Undergoing Bilateral Myringotomy and Placement of Ventilating Tubes
Brief Title: Postoperative Effects of Intranasal Fentanyl, IV and IM Morphine in Children Undergoing Myringotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Helena Karlberg, Associate Professor Department of Pediatrics and Anesthesiology Texas Children's Hospital Baylor College of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-21839
Record Dates: First submitted 2010-09-16; First posted 2010-11-19 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Otitis Media
Keywords: otitis media; recurrent ear infections (otitis media)
MeSH Terms: conditions — Otitis Media; Otitis | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IM morphine (Active Comparator): 0.1 mg/kg morphine IM
  Interventions: Drug: morphine IM
- IV morphine (Active Comparator): 0.1 mg/kg morphine IV
  Interventions: Drug: IV morphine
- fentanyl IN (Active Comparator): Intranasal fentanyl 2 mcg/kg IN
  Interventions: Drug: Intranasal fentanyl

INTERVENTIONS:
Drug: Intranasal fentanyl — 2mcg/kg fentanyl IN
  Arms: fentanyl IN
Drug: morphine IM — 0.1 mg/kg morphine IM for postop pain
  Arms: IM morphine
Drug: IV morphine — 0.1 mg/kg morphine IV
  Arms: IV morphine

SUMMARY:
The purpose of this study is to compare the difference in effect of three clinically common methods of providing pain medication during surgery for ventilating tubes placed for recurring ear infections.The methods are fentanyl dripped in the nose, morphine injected in a muscle, and morphine injected in a vein.

DETAILED DESCRIPTION:
Preoperative anxiety will be assessed by the modified Yale Preoperative Anxiety Scale (mYPAS) at two points - (1) prior to separating the patient from the caretaker and bringing the patient to the operating room and (2) on application of the facemask. In keeping with our current standard practice, the child will be brought to the OR without premedication, and anesthesia will be induced and maintained by having the child breath sevoflurane titrated up to 8 %, nitrous oxide 70 % and oxygen 30 % via a facemask. In keeping with the guidelines of the American Society of Anesthesiologists recommendations, standard monitoring of EKG, pulse oxymetry, blood pressure and skin temperature will be performed. After a satisfactory level of anesthesia has been achieved, intravenous access will be established. All patients will receive intranasal, IM and IV medications as assigned by a computer generated random number scheme.Group A -Intranasal Fentanyl 2 mcg/kg (0.04 ml/kg), Normal saline placebo IM and IV: Group B Intranasal normal saline (0.01 ml/kg) placebo, Morphine 0.1 mg/kg (0.01 ml/kg)IM and IV normal saline placebo (0.01 ml/kg); Group C- Intranasal Placebo - normal saline 0.04 ml/kg, IM normal saline Placebo 0.01 ml/kg and Morphine 0.1 mg/kg (0.01 ml/kg) IV.

The surgeon will be asked to describe the condition of the middle ear (worst side) on a scale of 1-4 as described by Davis et al. (1 = no fluid; 2 = serous fluid; 3 = pus; and 4 = thick tenacious mucus-glue ear). The surgeon will also report any laceration of the ear canal.

Induction time, surgery start and end time and arrival in PACU time will be recorded. In the postoperative care unit the pain score will be measured by the FLACC's pain scale (Face, Legs, Activity, Cry, Consolability), adverse emergence behavior will be measured by PAED scale described by Sikich et. al. (Pediatric Anesthesia Emergence Delirium Scale). Patients with pain scores greater than 4 will receive morphine 0.05 mg/kg IV, to be repeated once if the pain score remains greater than 4 after 10 minutes. Acetaminophen 10-15 mg/kg will be administered enterally for pain scores between 1-3.

The incidence of oxygen desaturation (pulse oximetry values less than 95% for greater than 30 secs), emesis and need for pain rescue medication will be recorded. The times of arrival in PACU, eye opening, response to command, ambulation, discharge readiness, and actual discharge home will be recorded as well. Parental satisfaction with postoperative pain control and the overall experience will be measured on a 10-point (0= completely dissatisfied -10= completely satisfied) verbal rating scale. A postoperative survey will be conducted over the phone the following day. Time and dose of postoperative medications, quality and duration of sleep, appetite and incidence of nausea and vomiting, time patient returned to presurgical level of playing and normal behavior and parent satisfaction will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* bilateral myringotomy

Exclusion Criteria:

* ASA greater than 2
* history of bleeding disorder/thrombocytopenia
* history of allergy to morphine or fentanyl

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Karlberg, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Result] Hippard HK, Govindan K, Friedman EM, Sulek M, Giannoni C, Larrier D, Minard CG, Watcha MF. Postoperative analgesic and behavioral effects of intranasal fentanyl, intravenous morphine, and intramuscular morphine in pediatric patients undergoing bilateral myringotomy and placement of ventilating tubes. Anesth Analg. 2012 Aug;115(2):356-63. doi: 10.1213/ANE.0b013e31825afef3. Epub 2012 Jun 5. PMID 22669347

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children scheduled for bilateral myringotomy and insertion of tubes at TCH from September 2008 to Feb 2011
Pre-assignment Details: 1531 children screened, 1143 excluded as not qualifying, 217 declined to participate
Period: Overall Study
Arm/Group | IM Morphine | IV Morphine | Fentanyl IN
Started | 59 | 55 | 57
Completed | 56 | 52 | 48
Not Completed | 3 | 3 | 9
Not completed — Protocol Violation | 3 | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IM Morphine | IV Morphine | Fentanyl IN | Total
Number analyzed (Participants) | 59 | 55 | 57 | 171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 59 | 55 | 57 | 171
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Limited to patients who completed study
  years | 2.3 (1.6) | 2.7 (2.2) | 2.4 (1.7) | 2.4 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 24 | 64
  Male | 36 | 38 | 33 | 107
Region of Enrollment [Number; unit: participants]
  United States | 59 | 55 | 57 | 171
Weight in Kgs [Mean (Standard Deviation); unit: Kgs] — Excluded 15 patients for protocol violations. These 15 patients did not undergo study procedures Baseline measures only of completed cases
  Kgs | 14.1 (7.3) | 15.2 (8.1) | 13.3 (4.6) | 14.2 (6.9)
Number completing study [Number; unit: participants] — 15 cases excluded for protocol violations including 3, 3 and 9 in the IM morphine, IV morphine and IN fentanyl groups respectively.
  participants | 56 | 52 | 48 | 156
Gender in patients completing study [Number; unit: Participants] — Excluding protocol violations
  Participants
    Male | 35 | 37 | 29 | 101
    Female | 21 | 15 | 19 | 55
ASA Physical Status in Patients who completed study [Number; unit: Participants] — Limited to those who completed study and excluding protocol violations
  ASA PHYSICAL STATUS CLASSIFICATION SYSTEM Last approved by the ASA House of Delegates on October 15, 2014 Definition ASA I A normal healthy patient Healthy, non-smoking, no or minimal alcohol use ASA II A patient with mild systemic disease Mild diseases only without substantive functional limitations.
  Participants
    ASA Physical Status 1 | 12 | 11 | 7 | 30
    ASA Physical Status 2 | 44 | 41 | 41 | 126

OUTCOME MEASURES:

1. Primary Outcome: Maximum Postoperative Face, Legs, Activity, Cry and Consolability (FLACC) Pain Score.
Description: FLACC assigns 0-2 points for each of 5 categories (face, legs, activity, cry, consolability)and sums these points to give a total score where high scores indicate worse pain (Paediatr Anaesth 2006; 16: 258-65)
Time Frame: Upon arrival in the PACU, and at 5, 10, 15, 30, 45, 60 minutes and at discharge
Population: Analysis was performed on per protocol basis excluding patients with protocol violations
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IM Morphine | IV Morphine | Fentanyl IN
Number analyzed (Participants) | 56 | 52 | 48
units on a scale | 2.9 (3.0) | 2.7 (3.2) | 2.0 (2.7)
Statistical Analysis 1: Comparison: IM Morphine vs IV Morphine vs Fentanyl IN; The primary outcome of the study was the maximum postoperative FLACC pain score; Test type: Superiority or Other; p = 0.21, Kruskal-Wallis; Kruskall Wallis ANOVA by ranks = 0.21, Standard Deviation 3.0

2. Secondary Outcome: Maximum PAED Score
Description: Maximum score on the Pediatric Anesthesia Emergence delirium scale. This has 5 items ranging from 1-4 and higher scores indicate greater emergence delirium.
  1. eye contact with care giver ,score 1-4, purposeful actions 1-4, aware of surrounding 1-4,restless 1-4, inconsolable 1-4, Maximum score 20.
Time Frame: Upon arrival in the PACU, and at 5, 10, 15, 30, 45, 60 minutes and at discharge
Population: The sample size was based on the assumption that the pain scores in the intranasal fentanyl group would be similar to those in previously published data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IM Morphine | IV Morphine | Fentanyl IN
Number analyzed (Participants) | 56 | 52 | 48
units on a scale | 6.1 (6.2) | 6.3 (6.7) | 4.6 (5.8)
Statistical Analysis 1: Comparison: IM Morphine vs IV Morphine vs Fentanyl IN; Kruskall Wallis test; Test type: Superiority or Other; p = 0.34, Kruskal-Wallis; Kruskall Wallis ANOVA = 0.34

ADVERSE EVENTS:
Arm/Group | IM Morphine | Fentanyl IN | IV Morphine
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 0/58 | 0/53 | 0/53

LIMITATIONS AND CAVEATS:
This study used an objective pain scale where the minimum clinically important difference in scores is unknown. The study did not use a group receiving no active treatment as this was unethical. We also did not measure blood levels of opioids.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No